CLINICAL TRIAL: NCT01620801
Title: A Phase 1 Safety Study in Subjects With Severe Hemophilia B (Factor IX Deficiency) Using a Single-Stranded, Adeno-Associated Pseudotype 8 Viral Vector to Deliver the Gene for Human Factor IX
Brief Title: Hemophilia B Gene Therapy With AAV8 Vector
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Collaborators: Children's Hospital of Philadelphia (Other); University of Pittsburgh (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAV8-hFIX19-101
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2018-12

CONDITIONS: Hemophilia B
Keywords: AAV; AAV8; Adeno-associated virus; Adeno-associated viral vectors; Hemophilia; Hemophilia B; Severe hemophilia B; Factor IX deficiency; Factor IX; FIX
MeSH Terms: conditions — Hemophilia B; Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose (Experimental): AAV8-hFIX19
  Interventions: Biological: AAV8-hFIX19
- Middle dose (Experimental): AAV8-hFIX19
  Interventions: Biological: AAV8-hFIX19
- High dose (Experimental): AAV8-hFIX19
  Interventions: Biological: AAV8-hFIX19

INTERVENTIONS:
Biological: AAV8-hFIX19 — One-time IV vector administration.

SUMMARY:
Hemophilia B is a bleeding disease in males due to very low levels of coagulation factor IX (FIX) in the blood. The current treatment is intravenous injection of FIX clotting factor concentrates, in response to bleeding. This study will focus on the severe, most common type of hemophilia B. This study plans to use a virus called adeno-associated virus (AAV), which in nature causes no disease, and can be engineered to deliver the human FIX gene (AAV8-hFIX19 vector) to liver cells, where FIX is normally made. This study will use the AAV8-hFIX19 vector.

DETAILED DESCRIPTION:
Hemophilia B is a bleeding disease in males due to very low levels of coagulation factor IX (FIX) in the blood. The major effect on health is joint disease caused by repeated bleeds into joints like the knee, hip, ankles and elbows. Rarely, the disease causes death due to bleeding into the brain or other important organs. The current treatment is intravenous injection of FIX clotting factor concentrates, in response to bleeding. This study will focus on the severe, most common type of hemophilia B.

This study plans to use a virus called adeno-associated virus (AAV), which in nature causes no disease, and can be engineered to deliver the human FIX gene (AAV8-hFIX19 vector) to liver cells, where FIX is normally made. Medical researchers in the United States and England have recently used an AAV vector similar to the one planned for this study, and found that after a single intravenous injection of the vector, blood levels of FIX reached levels greater than 1%, high enough to change the course of disease from severe to moderate. This means that the need to take FIX clotting factor concentrates has decreased, or even stopped. While these are important results, it needs to be noted that two of the six subjects who received the vector at higher doses developed inflammation of the liver. These subjects were treated with a steroid medication called Prednisolone, which is commonly used for serious types of inflammation. Prednisolone seemed to decrease the liver inflammation, as measured by a decrease in blood levels of elevated liver enzymes, and stability of FIX levels at greater than 1% of normal.

This study will use the AAV8-hFIX19 vector. The vector will be injected once into a peripheral vein of each subject, while the subject is in the hospital. If everything is fine, the subject will be discharged from the hospital the next day. Three doses of vector (low, middle, and high) will be tested in up to 15 different subjects, depending on safety outcome (as determined by blood and urine tests) and results of FIX levels. If some subjects develop liver inflammation, a short, tapering course of corticosteroids will be used.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to adhere to the clinical protocol and 15-year long-term follow-up as evidenced by written informed consent
* Adult males at least 18 years of age
* A. Severe FIX deficiency (<1% normal circulating FIX) or B. Moderately severe FIX deficiency (1-2% normal circulating FIX, inclusive) and a severe bleeding phenotype as defined by at least one of the following: i. On prophylaxis for a history of bleeding or ii. On demand therapy with a current or past history of frequent bleeding [4 or more bleeding episodes in the last 12 months or chronic hemophilic arthropathy (pain, joint destruction, and loss of range of motion) in one or more joints]
* No history of inhibitor against FIX
* No history of an allergic reaction or anaphylaxis to FIX products
* Greater than 20 exposure days of treatment with FIX protein
* Anti-AAV8 neutralizing titer measured at < 1:5
* Acceptable laboratory values: hemoglobin ≥ 11% gm; WBC ≥ 3,500/μL; platelets ≥ 100,000/μL; AST, ALT, alkaline phosphatase ≤ 2x ULN; bilirubin ≤ 1.2 gm/dL; and creatinine ≤ 1.5 gm/dL
* Subject agrees to use barrier contraception until at least two consecutive semen samples after vector administration are negative for vector sequences (may be for up to several months)

Exclusion Criteria:

* Subjects with active hepatitis B or C, and HBsAg or HCV RNA viral load positivity, respectively. Negative viral assays in two samples, collected at least six months apart, will be required to be considered negative. Both natural clearers and those who have cleared HCV on antiviral therapy are eligible.
* Subjects currently on antiviral therapy for hepatitis B or C
* Subjects with significant underlying liver disease, as defined by presence of portal hypertension, splenomegaly, varices, ascites, edema, gastrointestinal bleeding, encephalopathy, reduction below normal limits of serum albumin, or prior liver biopsy demonstrating significant fibrosis, specifically ≥ Metavir 3 fibrosis
* Subjects with serological evidence of HIV who have CD4 counts ≤ 200/mm3. Subjects who are HIV-positive and stable, with an adequate CD4 count (> 200/mm3) and undetectable viral load (< 50 gc/mL) measured twice in the six months prior to enrollment, on an antiretroviral drug regimen are eligible to enroll.
* History of inhibitor against FIX
* Anti-AAV8 antibody titers ≥ 1:5
* History of chronic infection or other chronic diseases which the investigators consider to constitute an unacceptable risk
* Subjects who have participated in a previous gene therapy research trial within one year of enrollment
* Subjects who have participated in a clinical study with an investigational drug within six months of enrollment
* Any other condition that would not allow the potential subject to complete follow-up examinations during the course of the study or, in the opinion of the investigator, makes the potential subject unsuitable for the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events related to investigational product | One year (with 15-year follow-up)
  Physical exams; clinical labs, including evaluation of FIX inhibitor; and adverse event reporting.

SECONDARY OUTCOMES:
Circulating plasma factor IX levels | One year (with 15-year follow-up)
  Factor IX activity and antigen; PT; and aPTT.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Spark Therapeutics, Inc.
Locations (3):
- United States (2):
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia